CLINICAL TRIAL: NCT03866967
Title: A Single-arm, Open-label, Multicenter Phase II Clinical Study of AK105 in Patients With Metastatic Nasopharyngeal Carcinoma After Failure of Second and Subsequent Lines of Chemotherapy
Brief Title: A Study of Anti-PD-1 AK105 in Patients With Metastatic Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: Akeso Tiancheng, Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK105-202
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: immunotherapy; Anti-PD-1 antibody; Nasopharyngeal Carcinoma; immuno-oncology
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AK105 (Experimental): Subjects receive AK105 200 mg intravenously (IV) once every 2 weeks (Q2W) until progression.
  Interventions: Biological: AK105

INTERVENTIONS:
Biological: AK105 — intravenous (IV) infusion

SUMMARY:
This is a multicenter, single-arm open-label, phase II study to evaluate the anti-tumor activity, safety, PK and immunogenicity of AK105 (Anti-PD1 antibody) in patients with metastatic nasopharyngeal carcinoma who have progressed after at least 2 prior lines of systemic chemotherapy (of which one of them must be platinum-based chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent form voluntarily.
* Age over 18 years old (inclusive) and not more than 75 years old (inclusive), when signing the ICF.
* Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.
* Expected life expectance ≥ 3 months.
* Histologically confirmed diagnosis of nonkeratinizing differentiated or undifferentiated NPC.
* Not suitable for radical local therapy.
* Stage IVb metastatic NPC patients who have failed the first-line platinum-based chemotherapy and the second-line chemotherapy.
* At least one measurable tumor lesion per RECIST 1.1 criteria. A lesion previously treated with local therapies such as radiotherapy can be considered a target lesion if there is objective evidence of progression in the lesion.
* Subjects must provide an available tumor tissue sample taken within 3 years prior to enrollment.
* Adequate organ function.
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception.
* Nonsterilized males who are sexually active with a female partner of childbearing potential must use highly effective method of contraception from Day 1 and for 120 days after the last dose of investigational product.

Exclusion Criteria:

* Receipt of last radiotherapy or any anti-tumor treatment [chemotherapy, targeted therapy, immunotherapy, Chinese herbal drugs with antitumor indications, or immunomodulators or tumor embolization] within 4 weeks prior to the first dose of study treatment. Nitrosourea or mitomycin C treatment within 6 weeks prior to the first dose of AK105.
* Prior exposure to any anti-PD-1, anti-PD-L1, anti-CTLA-4 antibody, or any other antibody or drug therapy for T cell co-stimulatory or checkpoint pathways, such as ICOS or agonists (e.g. CD40, CD137, GITR and OX40 etc).
* Other invasive malignancies within 2 years, except for locally treatable (manifested as cured) malignancies, such as basal or skin squamous cell carcinoma, superficial bladder cancer, cervical or breast carcinoma in situ.
* Subjects with active, known or suspected autoimmune disease, or a medical history of autoimmune disease, with the exceptions of the following: vitiligo, alopecia, Grave disease, psoriasis or eczema not requiring systemic treatment within the last 2 years, hypothyroidism (caused by autoimmune thyroiditis) only requiring steady doses of hormone replacement therapy and type I diabetes only requiring steady doses of insulin replacement therapy, or completely relieved childhood asthma that requires no intervention in adulthood, or primary diseases that will not relapse unless triggered by external factors.
* Active or previously documented inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis or chronic diarrhea).
* Subjects who require systemic corticosteroids (a dose equivalent to >10 mg/day prednisone) or other immunosuppressive drugs within 14 days prior to the first dose of study drug.
* Known history of testing positive for human immunodeficiency virus (HIV).
* Known history of primary immunodeficiency virus infection.
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* History of gastrointestinal perforation and/ or fistula within 6 months prior to enrollment.
* Necrotic lesion(s) found by examinations within 4 weeks prior to enrollment, which, in the investigator's opinion, is at risk of massive bleeding.
* Known history of interstitial lung disease.
* Known history of active tuberculosis (TB).
* Serious infections within 4 weeks prior to the first dose of study drug, including but not limited to complications requiring hospitalization, sepsis or severe pneumonia.
* An active infection requiring systemic therapy.
* Subjects with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) DNA exceeding 500 IU/ mL or active hepatitis C virus (HCV) should be excluded. Subjects with non-active HBsAg carriers, treated and stable hepatitis B (HBV DNA <500 IU/ mL) , and cured hepatitis C can be enrolled. Subjects with positive HCV antibodies are eligible only if the HCV RNA test results are negative.
* Major surgery (as defined by the investigator) within 30 days prior to the first dose of study drug.
* Presence of meningeal metastasis, spinal cord compression, leptomeningeal disease, or active brain metastasis.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
* Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v4.03 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria, with the exception of alopecia.
* Receipt of live or attenuated vaccination within 30 days prior to the first dose of study treatment, or plan to receive live or attenuated vaccine during the study.
* Known history of server hypersensitivity to other monoclonal antibodies.
* Known severe allergic reactions to paclitaxel, carboplatin, or their preventive medications.
* Known allergic reactions to any ingredients of AK105.
* Pregnant or lactating women.
* Any conditions that, in the investigator's opinion, may put subjects treated with the study drug at risks, or interfere with the evaluation of study drug or subject safety, or the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2021-03-13 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) assessed by IRRC per RECIST v1.1 for anti-tumor activity in the Full Analysis Set (FAS) population | up to 2 years
  ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) as assessed by IRRC and investigator | up to 2 years
  PFS is defined as the time from the date of randomization till the first documentation of disease progression (per RECIST v1.1 criteria) or death from any cause (whichever occurs first).
Disease control rate (DCR) as assessed by IRRC and investigator | up to 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD, based on RECIST v1.1.
Duration of response (DoR) as assessed by IRRC and investigator | up to 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | up to 2 years
  OS is defined as the time from the date of randomization to death from any cause.
Incidence and severity of treatment-emergent adverse events (TEAEs) | From the time of informed consent signed through 90 days after last dose of AK105
  An adverse event (AE) is any untoward medical occurrence or the deterioration of existing medical event in a clinical study subject administered an investigational drug, which does not necessarily have an unequivocal causal relationship with the investigational product.
Observed concentrations of AK105 | From first dose of AK105 through 90 days after last dose of AK105
  The endpoints for assessment of PK of AK105 include serum concentrations of AK105 at different timepoints after AK105 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK105 through 90 days after last dose of AK105
  The immunogenicity of AK105 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).
ORR as assessed by investigator per RECIST v1.1 for anti-tumor activity in the FAS population | up to 2 years
  ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.
Time to response (TTR) assessed by IRRC and investigator ； | up to 2 years
  TTR is defined as the time from the first dose of study drug to the first documented response (CR or PR).

CONTACTS AND LOCATIONS:
Overall Officials: Chaosu Hu, MD, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - FuDan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Z, Pang X, Zhong T, Qu T, Chen N, Ma S, He X, Xia D, Wang M, Xia M, Li B. Penpulimab, an Fc-Engineered IgG1 Anti-PD-1 Antibody, With Improved Efficacy and Low Incidence of Immune-Related Adverse Events. Front Immunol. 2022 Jun 27;13:924542. doi: 10.3389/fimmu.2022.924542. eCollection 2022. PMID 35833116
- See also: Related Info — https://www.nature.com/articles/s41392-024-01865-6